CLINICAL TRIAL: NCT00322686
Title: Efficacy and Safety of Oglemilast in the Prevention of Allergen-induced Bronchospasm
Brief Title: Study of Oglemilast for the Treatment of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: GRC-MD-03
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: oglemilast; asthma; allergen; prevention; prophylaxis; Allergen-Induced Asthma
MeSH Terms: conditions — Asthma | interventions — oglemilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oglemilast followed by placebo (Experimental)
  Interventions: Drug: Oglemilast
- Placebo followed by Oglemilast (Experimental)
  Interventions: Drug: Placebo then Oglemilast

INTERVENTIONS:
Drug: Oglemilast — Oglemilast, 15mg oral administration, once per day and then dose-matched placebo
  Arms: Oglemilast followed by placebo
Drug: Placebo then Oglemilast — Dose-matched placebo and then Oglemilast, 15mg, oral administration, once per day.
  Arms: Placebo followed by Oglemilast

SUMMARY:
The purpose of this study is to determine whether oglemilast is safe and effective in the treatment of allergen-induced asthma.

ELIGIBILITY:
Inclusion Criteria:

* Mild atopic asthma
* Hyperreactivity to methacholine
* Exhibit positive response to standard allergen skin prick test

Exclusion Criteria:

* Pulmonary disease other than asthma
* Asthma exacerbation within 4 weeks
* History of substance abuse
* Active cardiac disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of oglemilast in the prevention of bronchoconstriction after the administration of allergen, in comparison with placebo in patients with mild asthma | From Baseline to Day 7

SECONDARY OUTCOMES:
To evaluate the safety of oglemilast over 2 weeks as determined by adverse events,physical examinations, vital signs, electrocardiograms, and laboratory examinations | From Baseline to Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- Forest Investigative Site, Los Angeles, California, United States